CLINICAL TRIAL: NCT05243693
Title: Brentuximab Vedotin Plus Cisplatin, Cytarabine, and Dexamethasone in Patients With Relapsed or Refractory Hodgkin's Lymphoma Who Are Eligible for Transplant
Brief Title: Brentuximab Vedotin Plus DHAP in Relapsed or Refractory Hodgkin's Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Hyeon-Seok Eom, MD, PhD, Professor, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2020-0293
Record Dates: First submitted 2022-01-02; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Relapsed/Refractory Classical Hodgkin Lymphoma
MeSH Terms: conditions — Recurrence | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Brentuximab vedotin and DHAP (Experimental): A clinical study of safety and efficacy of treatment with Brentuximab vedotin and DHAP in patients with relapsed/refractory Hodgkin lymphoma
  Interventions: Drug: Brentuximab vedotin

INTERVENTIONS:
Drug: Brentuximab vedotin — 3 cycles of Brentuximab vedotin and DHAP
  Other Names: Adcetris

SUMMARY:
< STUDY DESIGN > This study is a multi-center phase II trial in patients with relapsed or refractory Hodgkin's lymphoma after first-line treatment.

< Treatment Schedule >

1. Induction phase

   * Patients who sign the informed consent form (ICF) receive BV-DHAP induction therapy within 21 days.
   * Tumor response is evaluated following 2 cycles of induction therapy. As a result of tumor response evaluation, PD (progressive disease) means a withdrawal from the study; and CR (complete response), PR (partial response), or SD (stable disease) requires peripheral blood stem cell collection (PBSCC) followed by additional one cycle of induction therapy.
   * Following a total of 3 cycles of induction therapy, tumor response is evaluated again. If the result turns out to be CR or PR, treatment goes on to autologous stem cell transplant (ASCT). SD or PD means a withdrawal from the study.
2. Consolidation phase - ASCT is performed in accordance with a protocol based on the relevant site's policy.

DETAILED DESCRIPTION:
< STUDY DESIGN > This study is a multi-center phase II trial in patients with relapsed or refractory Hodgkin's lymphoma after first-line treatment.

< Treatment Schedule >

1. Induction phase

   - Patients who sign the informed consent form (ICF) receive BV-DHAP induction therapy within 21 days.

   Study Drug Dosage will be as follows; Brentuximab vedotin: 1.8 mg/kg IV over 30 minutes D1 Cisplatin* 100 mg/m2 + NS 1000 mL CIV over 24 hours D1 Cytarabine* 2.0 g/m2 + 5% DW 250 mL IV over 3 hours twice a day D2 Dexamethasone 40 mg IV or PO D1-4

   *If baseline or on treatment creatinine clearance is less than 60 mL/min, 25% dose reduction should strongly be considered (cisplatin 75 mg/m2, cytarabine 1.5 g/m2)
   * Tumor response is evaluated following 2 cycles of induction therapy. As a result of tumor response evaluation, PD (progressive disease) means a withdrawal from the study; and CR (complete response), PR (partial response), or SD (stable disease) requires peripheral blood stem cell collection (PBSCC) followed by additional one cycle of induction therapy.
   * Following a total of 3 cycles of induction therapy, tumor response is evaluated again. If the result turns out to be CR or PR, treatment goes on to autologous stem cell transplant (ASCT). SD or PD means a withdrawal from the study.
   * Each cycle is implemented at an interval of 21 days (± 3 days).
2. Consolidation phase

   * ASCT is performed in accordance with a protocol based on the relevant site's policy.
   * Conditioning regimen will be determined by the attending physician. For example, BEAM, BuCyEtopo, BeEAM (Bendamustine+EAM), etc.
   * Other conservative managements will be carried out according to the policy of participating site

< Follow-Up Schedule >

* Patients will be recruited up to 3 years from the start date of this study.
* Primary analysis and reporting will be carried out at the completion of ASCT of the last patient.
* PFS and OS will be followed up for up to 2 years from the completion of ASCT of the last patient. Final analysis will be reported at this point.
* After completion of ASCT, a patient will be followed up at an interval of 3 months for 2 years

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of classical Hodgkin's lymphoma. CD30 has to be positive
2. Refractory to the first-line treatment or relapse after the first-line treatment (radiologically confirmed)

   * Deauville score 5 as a result of the restaging PET-CT after 2 to 3 cycles of ABVD treatment
   * Deauville score 4 to 5 even after the completion of ABVD treatment or radiotherapy and are not candidates for ISRT (involved site radiation therapy)
   * Radiologically confirmed relapsed after achieving CR
3. At least one measurable lesion(s)

   * nodal lesion longest transverse diameter (LDi) ≥ 1.5 cm
   * extranodal lesion LDi ≥ 1.0 cm)
4. Age 19 to 70 years
5. ECOG PS 0 - 2
6. Appropriate organ functions to tolerate the protocol treatment and ASCT Absolute Neutrophil Count (ANC) ≥ 1.5 x 10^9/L Platelets ≥ 75 x 10^9/L Hemoglobin ≥ 8.0 g/dL Serum Creatinine ≤ 1.5 x upper limit normal (ULN) Serum Bilirubin ≤ 1.5 x ULN AST and ALT ≤ 3 x ULN Corrected diffusing capacity for carbon monoxide (DLCO) ≥50 percent
7. Female patient is either post-menopausal for at least 1 year before the screening visit or surgically sterile or if of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 6 months after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse.
8. Male patients, even if surgically sterilized, (i.e., status post vasectomy) agree to practice effective barrier contraception during the entire study period and through 6 months after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse.
9. Written informed consent

Exclusion Criteria:

1. Non-Hodgkin's lymphoma or nodular lymphocyte predominant Hodgkin's lymphoma
2. 2 or more prior lines of treatment (Palliative radiotherapy or high-dose steroid therapy for symptom control are allowed)
3. Known cerebral or meningeal disease (HL or any other etiology), including signs or symptoms of PML
4. Confirmed CNS involvement and/or symptomatic neurologic disease compromising normal activities of daily living or requiring medications
5. Patients who cannot tolerate high-dose therapy followed by ASCT described in the inclusion criteria 6.
6. Patients with severe or uncontrolled medical conditions, abnormal laboratory findings, or psychiatric disorders. For example, i. severely impaired pulmonary function as defined as spirometry and DLCO (diffusing capacity of the lung for carbon monoxide) that is 50% or less of the normal predicted value and/or O2 saturation that is 90% or less at rest on room air ii. any active (acute or chronic) or uncontrolled infection/disorders that impair the ability to evaluate the patient or for the patient to complete the study iii. nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by this study drug, such as severe hypertension that is not controlled with medical management and thyroid abnormalities when thyroid function cannot be maintained in the normal range by medication iv. creatinine clearance < 30 mL/min
7. Known history of any of the following cardiovascular conditions i. Myocardial infarction within 2 years of enrollment ii. New York Heart Association (NYHA) Class III or IV heart failure iii. Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure (CHF), angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities iv. Recent evidence (within 6 months before first dose of study drug) of a left-ventricular ejection fraction <50%
8. Synchronous or metachronous malignant tumor other than HL within 5 years (except for adequately treated basal cell carcinoma (BCC) or squamous cell carcinoma (SCC) of the skin, carcinoma in situ of the uterine cervix, adequately resected differentiated thyroid cancer, intraepithelial carcinoma of the neck or breast, or prostate cancer that can be monitored for progress status without any treatment).
9. Hypersensitivity to the investigational products.
10. Peripheral neuropathy ≥ Grade 2
11. Pregnant or nursing women
12. Human immunodeficiency virus (HIV)-positive
13. Active hepatitis B or hepatitis C infection

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | up to 3 months
  Tumor response is evaluated following 3 cycles (each cycle is 21 days) of BV + DHAP induction therapy

SECONDARY OUTCOMES:
Progression free survival | up to 24 months
  PFS after BV + DHAP induction treatment & ASCT
Overall survival | up to 24 months
  PFS after BV + DHAP induction treatment & ASCT
Overall response rate | up to 3 months
  Tumor response is evaluated following 3 cycles (each cycle is 21 days) of BV+ DHAP induction therapy
Safety profiles | up to 3 months
  Frequency of grade 3 or higher treatment-related adverse events by CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon-Seok Eom, MD, PhD, Principal Investigator — National Cancer Center
Locations (1):
- Hyeon-Seok Eom, Goyang-si, Gyeonggi-do, South Korea